CLINICAL TRIAL: NCT04168580
Title: Brown Adipose Tissue as a Therapeutic for the Metabolic and Cardiac Dysfunction With Senescence (BATSR)
Acronym: BATSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1456947; R01AG060542 (NIH)
Record Dates: First submitted 2019-11-06; First posted 2019-11-19 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Diseases
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OA- Older Athlete (No Intervention): Older adults who are regularly engaged in endurance exercise
- OS- Older Sedentary (Active Comparator): Older adults who are sedentary
  Interventions: Other: Exercise Training Intervention

INTERVENTIONS:
Other: Exercise Training Intervention — Older sedentary participants will undergo 8 weeks of exercise training. The exercise program will be supervised by a certified exercise physiologist and will take place at the AdventHealth Translational Research Institute (TRI) exercise training facility. Exercise compliance will be monitored for exercise training 4 days per week (32 total sessions). Aerobic training will be 30 minutes of brisk walking, jogging, cycle ergometry. Walking will be the primary mode of aerobic exercise given its widespread popularity and ease of administration across a broad segment of the older adult population. Walking will be at a moderate intensity and determined based on Heart Rate (50-70% of Maximal Heart Rate from most recent VO2max) and rating of perceived exertion using Borg's scale (ranges from 6 to 20).
  Arms: OS- Older Sedentary

SUMMARY:
The goal of this study is to define the effect of aging on brown adipose tissue mass in a cohort of older sedentary and older athlete adults.

DETAILED DESCRIPTION:
Brown adipose tissue is a thermogenic tissue that contains large capacity to dissipate energy as heat. When activated by either cold-stimulation or increasing the amount of brown adipose tissue by transplantation, brown adipose tissue increases energy expenditure, decreases plasma glucose and lipids and improves systemic metabolism.

Brown adipose tissue has great potential as a therapeutic target to combat both metabolic and cardiovascular disease, but brown adipose tissue decreases with age. The objective of this study is to define the effect of aging on brown adipose tissue mass in a cohort of older sedentary and older athlete adults. Studying the role of brown adipose tissue will potentially help us understand and prevent an accelerated aging process, which will help researchers better understand metabolic and cardiac health in the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females between the ages of 65 to 90 years of age.
2. BMI 35kg/m2, inclusive at time of screening.
3. Stable weight (No gain/loss of ≥ 10 lbs within 6 months prior to screening).
4. Non-smokers as defined by not smoking any tobacco or using nicotine-containing products and not using vape pens or vaporizers within 3 months prior to screening.
5. Participant must have renal function with an estimated glomerular filtration rate (eGFR) > 45 ml/min/1.73m2 determined at screening.
6. Triglyceride level is < 350 mg/dl and LDL cholesterol is ≤ 150 mg/dl at screening.
7. States willingness to follow protocol as described, including the prescribed exercise level and completing any forms needed throughout the study.
8. Voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.

   Group Specific Inclusion Criteria:
9. Older Athletes (OA) Only: Endurance trained athletes, defined as exercising (running, cycling, swimming) >3days/wk for >6 months without layoff. This will be verified by self-report and triaxial accelerometry.
10. Older Sedentary (OS) Only: Defined as <1day/wk of structured exercise and determined by self-report and triaxial accelerometry.

Exclusion Criteria:

1. History of type 1 or type 2 diabetes per self-report at screening visit 1.
2. Actively pursuing weight loss and/or lifestyle changes at time of screening.
3. Untreated or poorly controlled hypertension (Systolic > 150, Diastolic > 95).
4. Mini Mental State Exam (MMSE) <21.
5. Participant has had a significant cardiovascular event (e.g. myocardial infarction, stroke) ≤ 6 months prior to screening visit; or stated history of congestive heart failure; or participant has evidence of cardiovascular disease assessed during the ECG at screening. In the event of a positive stress test, participants are referred to their primary care physician. If the electrocardiogram (ECG) is determined to be a false positive, participant may be allowed to participate in study after confirmatory records obtained.
6. Current infection (requiring prescription antimicrobial or antiviral medication, or hospitalization), or corticosteroid treatment (with the exception of inhaled or topical steroids) in the last 3 months prior to screening visit.
7. Participant is currently taking anti-inflammatory medication or has had anti-inflammatory medication within 1 week prior to screening (including over the counter formulations; e.g. Aleve, Motrin, ibuprofen, naproxen, low dose aspirin).
8. Surgery requiring >2 days of hospitalization in the last 3 weeks prior to screening visit.
9. Participant has an active malignancy (with the exception of basal cell) or autoimmune disease.
10. Participant has a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV, per self-report.
11. Participant is an amputee and/or has presence of partial or full artificial limb.
12. Participant currently has uncontrolled severe diarrhea, nausea or vomiting.
13. Participant has uncontrolled severe (including stage III or above) gastrointestinal absorption-related disorders, within 3 months of screening, such as: obstruction of the gastrointestinal tract, inflammatory bowel disease, short bowel syndrome, gastroesophageal reflux disease, gastroparesis, peptic ulcer disease, celiac disease, intestinal dysmotility, diverticulitis, ischemic colitis and bariatric surgery.
14. Cannot abstain from alcohol for the duration of the testing periods.
15. Subjects who fulfill any of the contraindications for MRI; examples include metal implants, devices, paramagnetic objects contained within the body and excessive or metal-containing tattoos.
16. Unable to participate in Magnetic Resonance or DEXA assessments due to physical limitations of equipment tolerances (e.g., MRI bore size and DEXA 450-pound weight limit), claustrophobia, or based on Investigator's judgment at screening.
17. Participant cannot refrain from taking medications/dietary supplements/herbals or substances that could modulate glucose metabolism, or are considered anabolic, or reduce weight (fat mass) in the opinion of the PI or Physician, starting two weeks prior to enrollment and over the entire course of the study. These include progestational agents, steroids, growth hormone, dronabinol, marijuana, calcium-betahydroxy-betamethylbutyrate (CaHMB), free amino acid supplements and dietary supplements to aid weight loss.
18. Participant has hypothyroidism (0.5mI U/L) or hyperthyroidism (10mI U/L).
19. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete the study.
20. Because all women participating in this project will be post-menopausal, there will be no need for a pregnancy test prior to DEXA procedures. Females currently on hormone replacement therapy can participate in the study if they have been on a stable dose of Hormone Replacement Therapy (HRT) for at least 6 months and will continue to be on HRT during the study.
21. Potential participants taking stable doses of medications for the last 30 days prior to screening for Blood pressure, cholesterol, gastroesophageal reflux disease (GERD) may be permitted to participate.
22. Participant becomes Covid-19 positive at any point during the study.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Coen, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OA- Older Athlete | OS- Older Sedentary
Started | 17 | 15
Completed | 15 | 15
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OA- Older Athlete | OS- Older Sedentary | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.47 (4.16) | 69.67 (3.99) | 69.57 (4.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Collection of Imaging of BAT by Magnetic Resonance Imaging
Description: Supraclavicular Adipose Tissue Proton Density Fat Fraction Percentage (PDFF %) is the primary outcome. PDFF % is determined by MRI
Time Frame: Baseline and 8 weeks (or Post-Exercise Training - for OS group only)
Population: The OA group did not complete the exercise training intervention and so there was no 8 week/post-exercise data collected for this group.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | OA- Older Athlete | OS- Older Sedentary
Number analyzed (Participants) | 15 | 15
Percentage
  Baseline | 78.69 (6.43) | 82.58 (7.28)
  Post-Exercise Training: number analyzed (Participants) | 0 | 15
  Post-Exercise Training |  | 82.45 (6.37)

2. Secondary Outcome: Aerobic Fitness
Description: As determine by a VO2max test
Time Frame: Baseline and 8 weeks (or Post-Exercise Training - for OS group only)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: VO2max (mL/min/kg)
Arm/Group | OA- Older Athlete | OS- Older Sedentary
Number analyzed (Participants) | 15 | 15
VO2max (mL/min/kg)
  Baseline | 30.4 (5.97) | 20.57 (4.39)
  Post Exercise Training: number analyzed (Participants) | 0 | 15
  Post Exercise Training |  | 20.71 (3.11)

3. Secondary Outcome: Body Composition
Description: Fat mass as determined by DEXA
Time Frame: Baseline and 8 weeks (or Post-Exercise Training - for OS group only)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | OA- Older Athlete | OS- Older Sedentary
Number analyzed (Participants) | 15 | 15
Kg
  Baseline | 19.23 (6.52) | 26.96 (8.57)
  Post Exercise Training: number analyzed (Participants) | 0 | 15
  Post Exercise Training |  | 26.63 (8.33)

4. Secondary Outcome: Muscle Testing - Power
Description: Right leg extension power as determined by Biodex (180deg/s)
Time Frame: Baseline and 8 weeks (or Post-Exercise Training - for OS group only)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Watt
Arm/Group | OA- Older Athlete | OS- Older Sedentary
Number analyzed (Participants) | 15 | 15
Watt
  Baseline | 127.7 (48.94) | 109.59 (41.83)
  Post Exercise Training: number analyzed (Participants) | 0 | 15
  Post Exercise Training |  | 107.99 (42.13)

ADVERSE EVENTS:
Time Frame: From Baseline to Week 8 (post exercise training) for the OS-Older Sedentary group only; and at Baseline for the OA-Older Athlete group.
Description: Study participants were assessed for AE occurrence at every study visit.
Arm/Group | OA- Older Athlete | OS- Older Sedentary
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 5/15 | 9/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OA- Older Athlete (N=15) | OS- Older Sedentary (N=15)
Runny nose, cough, sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nausea and Vomitting (Gastrointestinal disorders) | 1 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Left Arm Swelling at IV site (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
lateral epicondylitis (tennis elbow) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Issue with IV infiltration (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Benign Prostatic Hyperplasia (BPH) (Renal and urinary disorders) | 0 (0) | 1 (1)
Fall - Outside Study (not related to study) (Social circumstances) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT04168580/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT04168580/ICF_000.pdf